CLINICAL TRIAL: NCT01922635
Title: Validation of Metrological Properties of Questionnaire of Quality of Life LYMPHOQOL
Brief Title: Validation of Metrological Properties of Lymphoqol
Acronym: LYMPHOQOL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Modification the study with a new questionnaire was not successful.
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 8967
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Primary Lymhedema
Keywords: Primary lymphedema quality of life, genetic research

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Other: Valadation of the metrological properties of questionnaire of quality of life

INTERVENTIONS:
Other: Valadation of the metrological properties of questionnaire of quality of life

SUMMARY:
The constitutional lymphœdema is a rare disease with an annual incidence before the age of 20 years considered at 1,15/100 000. This chronic, incurable disease without hiring directly the prognosis for survival, alter the body image imposing a "visible" deformity and of which the treatment which aims at reducing and at stabilizing the physical deformation is binding and expensive. The lymphœdema is a crippling disease of the child. As such, it rings on the everyday life of the child and on the family environment. This question is all the more important, that all the studies show that the success of the treatment bases on the compliance in the concentration and in the care of hygiene. The parameters of the success of these treatments at the child are not known.

DETAILED DESCRIPTION:
In the literature we find no specific information on the psychic and social repercussions of the lymphœdema for the child who is affected. If the psychic and social repercussions of the secondary lymphœdema in the breast cancer are well known, very few things are it on those of the primary lymphœdema. Some studies estimate globally the quality of life of the patients with a lymphœdema whatever is the origin and the etiologie. These studies of money groups suggest that the psychic difficulties and of therapeutic care are not identical. A single study approaches the specific question of the lymphœdema of the child by focusing on the real-life experience of expanding child of a primary lymphœdema.The construction and the validation of a tool measuring the quality of life of the children and the young adults affected by lymphœdema congenital appears as a starting point. A tool which would first of all allow to make the current situation for the regional level, and then can envisage national actions common. According to recent studies, the evolution of the lymphoedema is different according to the forms of initial clinical expression of the lymphoedema, we wish we can thus know during this study the impact of these various clinical forms on the quality of life of the patients. A genetic collection will be realized for that purpose (genetic research).

ELIGIBILITY:
Inclusion Criteria:

* Primary lymphedema, stage 2 or 3 ISL

Exclusion Criteria:

* Primary lymphedema stage 1, secondary lymphedema, Minimum 6 years, maximum 25

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2013-07; Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Validation of the metrological properties of questionnaire of quality of life LYMPHOQOL | 3 Years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, Herault, France

REFERENCES:
- [Derived] Quere I, Stasi E, Mestre S, Roessler J, Roccatello D, Moffatt C. International Camps for Children with Lymphedema and Lymphatic Anomalies: When Education Links with Psychosocial Research. Lymphat Res Biol. 2021 Feb;19(1):36-40. doi: 10.1089/lrb.2020.0095. PMID 33625888